CLINICAL TRIAL: NCT04028739
Title: A Randomized, Open-label, Cross-over, Single Administration Study to Compare Bioavailability of Curcumin in Health Adults
Brief Title: Theracurmin vs Curcumin Bioavailability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TC_BA
Record Dates: First submitted 2019-07-17; First posted 2019-07-23 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Bioavailability
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Theracurmin CR-033P (Experimental): 1 Capsule with 150mL water, Single, curcumin 90mg/day
  Interventions: Dietary Supplement: curmin
- Theracurmin CR-031P (Experimental): 3 Capsule with 150mL water, Single, curcumin 90mg/day
  Interventions: Dietary Supplement: curmin
- Curcumin (Experimental): 1 Capsule with 150mL water, Single, curcumin 90mg/day
  Interventions: Dietary Supplement: curmin

INTERVENTIONS:
Dietary Supplement: curmin — curcumin 90mg/day cross-over
  Other Names: Theracurmin CR-033P; Theracurmin CR-031P; Curcumin

SUMMARY:
A randomized, open-label, cross-over, single administration study to compare bioavailability of curcumin in health adults

DETAILED DESCRIPTION:
* Randomization, Open-label, 3-period, 6-sequence, Crossover, Single
* Drug-free inverval : more than 7 days
* Sampling time : 0,0.5,1,1.5,2,3,4,6,8,12h

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult 19 to 60 years
2. BMI 18.0~30.0kg/m2 at screening
3. Subject who was given, and fully understood, the information about the study, and has provided voluntary written informed consent to participate in the study and agreed to comply with the study requirements.

Exclusion Criteria

1. A person with clinically significant disease corresponding to cardiovascular, respiratory, liver, kidney, digestive system, blood/tumor system, endocrine system, immune system, neuropsychiatry or who has a history within the last 6 months.
2. A person with a history of gastrointestinal disease or surgery (except for simple cecal surgery or hernia surgery) that may affect the absorption of food for clinical research.
3. Persons who have an irritable reaction to foods containing turmeric or other drugs and food.
4. Those who took medicines within 7 days before the first intake of food for clinical research.
5. Food for Clinical Research If you have consumed foods containing turmeric (eg, radishes, curry) within 7 days before the first intake of food, or you can't consume until the day of intake of food for the last clinical study.
6. Those who have participated in other clinical studies within 90 days prior to the first intake of food for clinical research.
7. Women who are pregnant or lactating during screening, or who plan to become pregnant during clinical research. A person who is deemed unsuitable for participating in this clinical study because of other reasons.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Cmax | 12hours
  Maximum concentration at steady state
AUC | 12hours
  Area under the concentration-time curve at steady state

CONTACTS AND LOCATIONS:
Overall Officials: Hyewon Chung, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea Kuro Hospital, Seoul, South Korea